CLINICAL TRIAL: NCT04118881
Title: Preoperative Ear Acupuncture to Prevent Delayed Gastric Emptying After Pancreatoduodenectomy.A Single-center Prospective Randomized Controlled Clinical Study.
Brief Title: Ear Acupuncture Preventing Delayed Gastric Emptying.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E2019158A
Record Dates: First submitted 2019-09-26; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-08

CONDITIONS: Auricular Acupoint Embedding; Pancreaticoduodenectomy; Delayed Gastric Emptying
MeSH Terms: conditions — Gastroparesis | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): The treatment group was given intradermal needling at ear acupoints: cardia (CO3), stomach (CO4), sympathetic (HX4)
  Interventions: Other: Ear Acupuncture
- control group (Sham Comparator): The control group was given intradermal needling at ear acupoints: spiral area (HX7 and HX8).
  Interventions: Other: Ear Acupuncture

INTERVENTIONS:
Other: Ear Acupuncture — Auricular Acupuncture (AA) is a micro-system of acupuncture and moxibustion initiated by Chinese and French doctors. All acupoints are distributed in the ear. In the treatment of perioperative patients, ear needle is far away from the surgical wound and its minimally invasive and tolerable position has obvious advantages over body needle.AA can regulate the function of corresponding organs at acupoints. The theoretical basis of TCM is holistic concept and syndrome differentiation and treatment.AA can prevent and treat perioperative nausea and vomiting. A number of randomized controlled trials and retrospective studies have confirmed that AA has obvious advantages in preventing nausea and vomiting in perioperative period compared with routine prevention, and its possible mechanism is ear-directed stimulation of the ear branch of vagus nerve, thereby enhancing gastrointestinal motility and accelerating gastric emptying.

SUMMARY:
Pancreatoduodenectomy is the preferred surgical method for periampullary diseases. The most common complication is gastric emptying disorder, which often greatly affects the quality of life of patients and prolongs the length of hospitalization. There are few reports on the treatment of gastric emptying disorder with single method, poor continuity of curative effect and low level of evidence. This study is to explore the clinical efficacy and safety of ear acupuncture in the prevention and treatment of DGE after pancreaticoduodenal surgery. This study is divided into two parts. The first part is to study the clinical efficacy and safety of auricular acupoint embedding in preventing gastric emptying disorder after pancreaticoduodenectomy. The second part is to study the clinical efficacy and safety of electroacupuncture in treating gastric emptying disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent pancreaticoduodenectomy;
* No delayed gastric emptying or gastrointestinal obstruction before operation.
* ECOG score 0-2;
* No opioid analgesia or gastrointestinal motility drugs were administered for more than one week before operation.
* Adequate blood cell counts were available during the screening period.
* The blood biochemical indexes during screening period were as follows (48 hours before operation to 14 days before operation): AST (SGOT), ALT (SGPT) were less than or equal to the upper limit of 2.5 times normal value (ULN). Total bilirubin is less than or equal to 300 micromol/L. ULN serum creatinine is within the normal limit, or the level of serum creatinine is higher or lower than the normal value of institutions, but the calculated clearance rate is greater than or equal to 60 mL/min/1.73 m2. If the creatinine clearance rate is used, the actual body weight should be used to calculate the creatinine clearance rate (e.g. using the Cockroft-Gault formula).
* Coagulation function is normal.
* Male or non-pregnant and non-lactating women who were older than or equal to 18 years old signed the informed consent. If a female patient is of childbearing age (regular menstrual proof), the pregnancy test (such as serum beta-hCG) before the first study of drug administration must be negative. If patients are sexually active, they must agree to use contraceptive methods that researchers believe are adequate and appropriate during the study of drug administration. In addition, male and female patients must take contraceptive measures after treatment, as recommended by the product prescription information provided in the study manual.
* The patient has been informed of the nature of the study and has agreed to participate in the study and signed an informed consent before participating in any research-related activities.
* Ability to comply with research visits and other programme requirements

Exclusion Criteria:

* The patient did not receive standard pancreaticoduodenectomy.
* Myocardial infarction, severe or unstable angina pectoris, coronary artery or peripheral artery bypass grafting, New York Heart Association (NYHA) grade III-IV heart failure, cerebrovascular accident, transient ischemic attack or epileptic seizure occurred within 30 days before operation.
* Any condition that may impair patient safety or the integrity of research data, including serious medical risk factors, medical events, laboratory abnormalities or psychiatric disorders;
* The patient's access to any other clinical study or to a trial of an interventional drug may interfere with the evaluation of this study procedure.
* Patients are unwilling or unable to follow the research procedure;
* Researchers do not think it is suitable for inclusion.
* Acupuncture and moxibustion is currently used or used in the past 30 days.
* Ear trauma or unhealed ear wound
* Stainless steel allergists

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-10-10 (Estimated); Primary Completion 2021-08-02 (Estimated); Study Completion 2021-12-02 (Estimated)

PRIMARY OUTCOMES:
Grading of delayed gastric emptying | Day3 after operation
  The assessment was conducted in accordance with the DGE guidelines for post-PD surgery issued by the International Research Group of Pancreatic Surgery (ISGPS) in 2007.
Grading of delayed gastric emptying | Day5 after operation
  The assessment was conducted in accordance with the DGE guidelines for post-PD surgery issued by the International Research Group of Pancreatic Surgery (ISGPS) in 2007.
Grading of delayed gastric emptying | Day7 after operation
  The assessment was conducted in accordance with the DGE guidelines for post-PD surgery issued by the International Research Group of Pancreatic Surgery (ISGPS) in 2007.
Grading of delayed gastric emptying | Day14 after operation
  The assessment was conducted in accordance with the DGE guidelines for post-PD surgery issued by the International Research Group of Pancreatic Surgery (ISGPS) in 2007.

SECONDARY OUTCOMES:
Changes of motilin before and after operation | Day0 and Day7 after operation.
  Serum motilin was measured at Day0 and Day7 after operation.
Changes of somatostatin before and after operation | Day0 and Day7 after operation.
  Somatostatin were measured at Day0 and Day7 after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China